CLINICAL TRIAL: NCT03187197
Title: Patients Assessment of Satisfaction for Stroke Prevention in Atrial Fibrillation Impact of Conventional Oral Anticoagulant (OAC) Compared With Novel Oral Anticoagulant (NOAC)
Brief Title: Patients' Assessment of Satisfaction for Stroke Prevention in Atrial Fibrillation
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1160-0286
Record Dates: First submitted 2017-06-13; First posted 2017-06-14 (Actual); Results first posted 2020-02-24 (Actual); Last update posted 2020-02-24 (Actual); Status verified 2020-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort A: consented patients with NVAF in Taiwan with a previous VKA therapy, followed by switching to Pradaxa®
  Interventions: Drug: Pradaxa®
- Cohort B: patients being newly diagnosed with NVAF and initiated on Pradaxa®
  Interventions: Drug: Pradaxa®

INTERVENTIONS:
Drug: Pradaxa® — Dabigatran etexilate
  Other Names: Dabigatran etexilate

SUMMARY:
To describe the treatment perception from patients with non-valvular atrial fibrillation (NVAF) receiving Pradaxa® or VKA for stroke prevention by using the self-estimation questionnaire of PACT-Q during a 6-month study period.

ELIGIBILITY:
Inclusion criteria:

Cohort A (patients switched from VKA to Pradaxa)

* Written informed consent prior to participation.
* Female or male patients ≥ 20 years of age with a diagnosis of non-valvular atrial fibrillation (NVAF).
* At least 3 months of continuous VKA treatment for stroke prevention prior to baseline assessment.
* Patients switched to Pradaxa prior to baseline assessment according to the physician's discretion and the Summary of Product Characteristics (SmPCs)/reimbursement criteria.

OR Cohort B (patients newly initiated Pradaxa or VKA)

* Written informed consent prior to participation.
* Female or male patients ≥ 20 years of age, newly diagnosed with NVAF, and no previous treatment for stroke prevention (no use of any OAC within 1 year prior to enrolment).
* Patients initiated stroke prevention treatment with Pradaxa or VKA according to the physician's discretion and the SmPCs/reimbursement criteria.

Exclusion criteria:

* Contraindication to the use of Pradaxa® or VKA as described in the SmPCs.
* Patients receiving Pradaxa® or VKA for any other condition than stroke prevention in NVAF.
* Current participation in any clinical trial of a drug or device.
* Current participation in an AF-related registry, e.g. the Gloria AF program.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 20 years of age or older with a diagnosis of non-valvular atrial fibrillation (NVAF).
Sampling Method: Non-Probability Sample
Enrollment: 1315 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (24):
- Taiwan (24):
  - Chang-Hua Christian Hospital, Changhua
  - Show Chwan Memorial Hospital, Changhua
  - Chia-Yi Christian Hospital, Chia-Yi City
  - Hsinchu MacKay Memorial Hospital, Hsinchu
  - National Taiwan University Hospital-Hsin-Chu Branch, Hsinchu
  - Kaohsiung Medical University Chung-Ho Memorial Hospital, Kaohsiung City
  - E-Da Hospital, Kaohsiung City
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Medical University-Shuang Ho Hospital, New Taipei City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - NCKUH, Tainan
  - Chi Mei Medical Center, Tainan
  - Tainan Municipal An-Nan Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipe Veterans General Hospital, Taipei
  - Tri-Service General Hospital, Taipei
  - Shin Kong International HealthCare Center, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Chang Gung Memorial Hospital(TaoYuan), Taoyuan District
  - National Taiwan University Hospital Yun-Lin Branch, Yunlin County

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CW, Liu ME, Lee TM, Chang RY, Huang CY, Hu YF, Yeh HI. Patient satisfaction with dabigatrean and warfarin for stroke prevention in atrial fibrillation: Taiwan PASSION study. J Chin Med Assoc. 2021 Apr 1;84(4):375-382. doi: 10.1097/JCMA.0000000000000496. PMID 33784265

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study enrolled patients in Taiwan with a previous Vitamin K Antagonist (VKA) therapy, followed by switching to Pradaxa® (one of the novel oral anticoagulants (NOACs)) or patients being newly diagnosed with Non-Valvular Atrial Fibrillation (NVAF) and initiated on Pradaxa® or VKA.
Pre-assignment Details: Data was collected from approximately 20 medical centers or regional hospitals in Taiwan where Pradaxa® is taken as the prescription of stroke prophylaxis (or prevention) in Atrial Fibrillation (AF). Data was collected between June 23, 2017 and Jan 11, 2019. 10 enrolled participants were removed due to screening failures before entering the study.
Groups:
- Cohort A: Patients with a diagnosis of NVAF, who were using VKA therapy for at least 3 months for stroke prevention before entering the study and were switched to Pradaxa®, received 110 or 150 milligram (mg) Pradaxa® capsules twice daily.
- Cohort B - Pradaxa®: Patients newly diagnosed with NVAF, not previously treated with an anticoagulant for the prevention of stroke and initiated 110 or 150 mg Pradaxa® capsules twice daily.
- Cohort B - VKA: Patients newly diagnosed with NVAF, not previously treated with an anticoagulant for the prevention of stroke, and initiated VKA therapy. The choice of VKA and the appropriate dosing was at the discretion of the physician.
Period: Overall Study
Arm/Group | Cohort A | Cohort B - Pradaxa® | Cohort B - VKA
Started (Started are Enrolled) | 153 | 1097 | 55
Started (Eligible Participants as FAS) | 139 | 1052 | 54
Completed | 107 | 704 | 32
Not Completed | 46 | 393 | 23
Not completed — Stopped Pradaxa®/VKA | 11 | 65 | 4
Not completed — Withdrawal by Subject | 8 | 63 | 4
Not completed — Lost to Follow-up | 1 | 60 | 7
Not completed — Adverse Event | 6 | 29 | 0
Not completed — Death | 0 | 11 | 0
Not completed — Administrative problem | 1 | 1 | 0
Not completed — Reason not listed | 2 | 54 | 1
Not completed — Missing | 1 | 32 | 3
Not completed — Status missing | 2 | 33 | 3
Not completed — NA in incl/excl criteria, not analyzed. | 14 | 45 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): This set included all subjects who were eligible for study participation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort A | Cohort B - Pradaxa® | Cohort B - VKA | Total
Number analyzed (Participants) | 139 | 1052 | 54 | 1245
Age, Continuous [Mean (Standard Deviation); unit: Years] | 68.4 (15.65) | 71.5 (13.08) | 67.1 (12.88) | 71.0 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 431 | 17 | 505
  Male | 82 | 621 | 37 | 740
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 139 | 1052 | 54 | 1245
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 139 | 1052 | 54 | 1245
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 0 | 0
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Mean Perception of Anticoagulant Treatment Questionnaire 2 (PACT-Q2) Scores, for Patients in Cohort A, at Second and Last Assessment Compared to Baseline Assessment
Description: The PACT-Q was a self-administered questionnaire which was developed as a means to investigate patients´ satisfaction with anticoagulant treatment and treatment convenience in patients with deep venous thrombosis (DVT), pulmonary embolism (PE) or atrial fibrillation (AF). The PACT-Q2 was composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). Items for convenience and for burden of disease and treatment were reversed(reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score (CDS). Items for anticoagulant treatment satisfaction were summed and rescaled on a 0-100 scale to determine the satisfaction dimension score (SDS). High scores were more favorable. The two dimension scores were presented for Baseline, Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: Baseline, Visit 2 (30-45 days after initiation on Pradaxa®), Visit 3 (150-210 days after initiation on Pradaxa®).
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cohort A
Number analyzed (Participants) | 139
Units on Scale
  Convenience - Baseline: number analyzed (Participants) | 136
  Convenience - Baseline | 86.9 (13.31)
  Convenience - Visit 2: number analyzed (Participants) | 133
  Convenience - Visit 2 | 91.7 (10.74)
  Convenience - Visit 3: number analyzed (Participants) | 107
  Convenience - Visit 3 | 95.2 (6.48)
  Satisfaction - Baseline: number analyzed (Participants) | 138
  Satisfaction - Baseline | 64.3 (11.06)
  Satisfaction - Visit 2: number analyzed (Participants) | 135
  Satisfaction - Visit 2 | 68.1 (13.36)
  Satisfaction - Visit 3: number analyzed (Participants) | 107
  Satisfaction - Visit 3 | 72.5 (12.41)
Statistical Analysis 1: Comparison: Cohort A; Within group comparison of Baseline convenience with that of Visit 2; Test type: Other; p = 0.0001, Paired t-test
Statistical Analysis 2: Comparison: Cohort A; Within group comparison of Baseline convenience with that of Visit 3; Test type: Other; p = 0.0001, Paired t-test
Statistical Analysis 3: Comparison: Cohort A; Within group comparison of Baseline satisfaction with that of Visit 2; Test type: Other; p = 0.0031, Paired t-test
Statistical Analysis 4: Comparison: Cohort A; Within group comparison of Baseline satisfaction with that of Visit 3; Test type: Other; p = 0.0001, Paired t-test

2. Primary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort B, at Second and Last Assessment Compared Between Treatment Groups
Description: The PACT-Q2 was composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). The PACT-Q2 was to be administered to patients once treatment was ongoing. Items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction were summed and rescaled on a 0-100 scale to determine the satisfaction dimension score. High scores were more favorable. The two dimension scores were presented for Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD). Propensity score matching (PSM) method was used to identify matched Pradaxa® and VKA patients. Only the matched patients in each treatment group was summarized and used for comparison.
Time Frame: Visit 2 (30-45 days after initiation on Pradaxa® or VKA) and Visit 3 (150-210 days after initiation on Pradaxa® or VKA).
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Cohort B - Pradaxa® | Cohort B - VKA
Number analyzed (Participants) | 1052 | 54
Units on Scale
  Pre-PSM Convenience - Visit 2: number analyzed (Participants) | 926 | 47
  Pre-PSM Convenience - Visit 2 | 92.4 (9.88) | 94.3 (5.61)
  Pre-PSM Convenience - Visit 3: number analyzed (Participants) | 716 | 34
  Pre-PSM Convenience - Visit 3 | 93.9 (8.41) | 94.3 (6.35)
  Pre-PSM Satisfaction - Visit 2: number analyzed (Participants) | 931 | 47
  Pre-PSM Satisfaction - Visit 2 | 70.1 (11.51) | 67.3 (9.17)
  Pre-PSM Satisfaction - Visit 3: number analyzed (Participants) | 718 | 34
  Pre-PSM Satisfaction - Visit 3 | 73.9 (12.05) | 75.1 (11.95)
  PSM Convenience - Visit 2: number analyzed (Participants) | 2 | 2
  PSM Convenience - Visit 2 | 98.5 (2.18) | 80.8 (9.79)
  PSM Satisfaction - Visit 2: number analyzed (Participants) | 2 | 2
  PSM Satisfaction - Visit 2 | 71.4 (0.00) | 64.3 (2.02)
Statistical Analysis 1: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 2 treatment convenience before PSM; Test type: Other; p = 0.7879, t-test, 2 sided
Statistical Analysis 2: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 3 treatment convenience before PSM; Test type: Other; p = 0.6110, t-test, 2 sided
Statistical Analysis 3: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 2 treatment satisfaction before PSM; Test type: Other; p = 0.0832, t-test, 2 sided
Statistical Analysis 4: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 3 treatment satisfaction before PSM; Test type: Other; p = 0.6488, t-test, 2 sided
Statistical Analysis 5: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 2 treatment convenience after PSM; Test type: Other; p = 0.1301, Two sample T test
Statistical Analysis 6: Comparison: Cohort B - Pradaxa® vs Cohort B - VKA; Between group comparison of Visit 2 treatment satisfaction after PSM; Test type: Other; p = 0.1257, Two sample T test

3. Secondary Outcome: Mean PACT-Q2 Scores, for Patients in Cohort A, at Last Assessment Compared to Second Assessment
Description: The PACT-Q2 was composed of three dimensions covering: convenience (11 items), burden of disease and treatment (2 items), and anticoagulant treatment satisfaction (7 items). The PACT-Q2 was to be administered to patients once treatment was ongoing. Items for convenience and for burden of disease and treatment were reversed (reversed score = 6 - item score), added together and rescaled on a 0-100 scale to obtain the convenience dimension score. Items for anticoagulant treatment satisfaction were summed and rescaled on a 0-100 scale to determine the satisfaction dimension score. High scores were more favorable. The two dimension scores were presented for Visit 2 (second assessment) and Visit 3 (last assessment) as mean and standard deviation (SD).
Time Frame: Visit 2 (30-45 days after initiation on Pradaxa®) and Visit 3 (150-210 days after initiation on Pradaxa®).
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Cohort A
Number analyzed (Participants) | 139
Units on scale
  Convenience - Visit 2: number analyzed (Participants) | 133
  Convenience - Visit 2 | 91.7 (10.74)
  Convenience - Visit 3: number analyzed (Participants) | 107
  Convenience - Visit 3 | 95.2 (6.48)
  Satisfaction - Visit 2: number analyzed (Participants) | 135
  Satisfaction - Visit 2 | 68.1 (13.36)
  Satisfaction - Visit 3: number analyzed (Participants) | 107
  Satisfaction - Visit 3 | 72.5 (12.41)

4. Secondary Outcome: Description of PACT-Q1 Items for Patients in Cohort B at Baseline
Description: The PACT-Q1 was composed of a single dimension (7 items), covering the expectations of patients regarding their anticoagulant treatment, and was to be administered before treatment initiation. The 7 items were: Q1: How confident are you that your anticoagulant treatment will prevent blood clots? Q2: Do you expect that your anticoagulant treatment will relieve some of the symptoms you experience? Q3: Do you expect that your anticoagulant treatment will cause side effects such as minor bruises or bleeding? Q4: How important is it for you to have an anticoagulant treatment that is easy to take? Q5: How concerned are you about making mistakes when taking your anticoagulant treatment? Q6: How important is it for you to take care of your anticoagulant treatment by yourself? Q7: How concerned are you about how much you pay for your anticoagulant treatment? Responses ranged from 1 (Not at all) to 5 (Extremely/Completely/Very much).
Time Frame: Baseline
Population: FAS
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Cohort B - Pradaxa® | Cohort B - VKA
Number analyzed (Participants) | 1052 | 54
Units on scale
  Q1: number analyzed (Participants) | 1047 | 54
  Q1 | 3.2 (1.13) | 3.0 (0.99)
  Q2: number analyzed (Participants) | 1050 | 54
  Q2 | 3.2 (1.19) | 3.1 (1.11)
  Q3: number analyzed (Participants) | 1049 | 54
  Q3 | 2.3 (1.09) | 2.1 (1.00)
  Q4: number analyzed (Participants) | 1049 | 54
  Q4 | 3.6 (1.15) | 3.7 (1.21)
  Q5: number analyzed (Participants) | 1048 | 54
  Q5 | 2.8 (1.42) | 2.7 (1.54)
  Q6: number analyzed (Participants) | 1049 | 54
  Q6 | 3.7 (1.12) | 3.7 (1.09)
  Q7: number analyzed (Participants) | 1048 | 54
  Q7 | 2.4 (1.39) | 1.9 (1.21)

ADVERSE EVENTS:
Time Frame: From signing the informed consent till end of the study; up to 210 days.
Description: For AE reporting the safety set included all enrolled subjects with at least one actual follow-up.
  Following the updated Guidelines, the cardiologists treat participants using NOAC rather than VKA.
  There is a a major difference of patients included in the various cohorts ; this can be explained by the fact that it is a non-interventional, observational study. Which kind of treatment patients received was based on the investigators' decision according to the patient clinical situation.
Arm/Group | Cohort A | Cohort B - Pradaxa® | Cohort B - VKA
All-Cause Mortality (participants affected / at risk) | 0/148 | 11/978 | 0/48
Serious Adverse Events (participants affected / at risk) | 1/148 | 4/978 | 0/48
Other Adverse Events (participants affected / at risk) | 0/148 | 0/978 | 0/48
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort A (N=148) | Cohort B - Pradaxa® (N=978) | Cohort B - VKA (N=48)
Embolic stroke (Nervous system disorders) | 1 | 0 | 0
Septic shock (Infections and infestations) | 0 | 1 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Death (General disorders) | 0 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-18): https://cdn.clinicaltrials.gov/large-docs/97/NCT03187197/SAP_000.pdf
  • Study Protocol (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/97/NCT03187197/Prot_001.pdf